CLINICAL TRIAL: NCT06419790
Title: Effect of Electrode Belt Used for Lung Monitoring With Electrical Impedance Tomography on Tidal Volume of Healthy Volunteers
Brief Title: Effect of Electrode Belt Used for Lung Monitoring With EIT on Tidal Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: C3/017
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: EIT Electrode Belt Stiffness; Tidal Volume Changes
Keywords: electrode belt; EIT; spirometry; tidal volume
MeSH Terms: interventions — Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): Data were obtained at two phases at supine semi-sitting position during 15 min sponatenous breathing and 1 min forced breathing. Subjects were breathing through spirometric probe first without electrode belt, and second with electrode belt placed tightly around the thorax as recommened by the manufacturer.
  Interventions: Device: EIT electrode belt, spirometry

INTERVENTIONS:
Device: EIT electrode belt, spirometry — Placing electrode belt for EIT monitoring and measuring tidal volume with spirometer

SUMMARY:
Tidal volumes of ten spontaneously breathing healthy volunteers were measured using spirometer in two situations: wearing EIT electrode belt and without electrode belt. The changes of the tidal volumes were analysed in order to conclude whether the electrode belt has any impact on the volumes.

DETAILED DESCRIPTION:
Ten healthy, spontaneously breathing volunteers were in supine semi-sitting position and their tidal volume was measured for 15 min using spirometer Ergostick (Geratherm) twice: with electrode belt placed around the subjcest thorax in the level of 4th to 6th intercostal space in the parasternal line, and then without the electrode belt. The subjects were breathing for approx. 15 min sponatenously with deep, forced breathing in the last minute.

The stiff silicone electrode belt used for lung monitoring with electrical impedance tomography system PulmoVista 500 (Dräger Medical) is being placed tightly around the subjects chest in order to monitor distribution of the ventilation. The aim of the study is to analyse the differences in tidal volumes of the spontaneously breathing subject with and without the electrode belt.

Since the electrode belt is relatively stiff and the manufacturer recommends putting the belt on tightly, there is a possibility that it affects the breathing effort of the spontaneously breathing patients, which could possibly lead to lower tidal volumes.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* morbid obesity
* Tiffeneau index lower than 80 %
* wounded skin in the electrode belt location

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in tidal volumes | 15 minutes
  Analysing the changes of tidal volumes caused by the presence of electrode belt

CONTACTS AND LOCATIONS:
Overall Officials: Kristýna Koldová, Ph.D., Study Director — Faculty of Biomedical Engineering, Czech Technical University in Prague
Locations (1):
- Faculty of Biomedical Engineering, Czech Technical University in Prague, Kladno, Czechia

IPD SHARING:
Plan to Share IPD: No